CLINICAL TRIAL: NCT06091774
Title: Klinische Studie Zur Untersuchung Und Validierung Eines Therapieverfahrens Zur Einstellung Von Risikofaktoren Bei Patienten Mit Koronarer Herzkrankheit (KHK) Mittels Digitaler Therapiesteuerung
Brief Title: Clinical Study for the Investigation and Validation of a Therapy Procedure for the Adjustment of Risk Factors in Patients With Coronary Heart Disease by Means of Digital Therapy Control
Acronym: ERKHA
Status: Recruiting | Type: Observational
Sponsor: iATROS GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: 03
Record Dates: First submitted 2023-09-29; First posted 2023-10-19 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Coronary Artery Disease; Cardiovascular Diseases; Coronary Heart Disease; Ischemic Heart Disease
Keywords: eHealth; cardiology; coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease; Cardiovascular Diseases; Coronary Disease; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group with the medical device "iATROS": Patients are subsequently assigned to one of the two groups in a 1:1 randomization.
  The treatment to be carried out in the intervention group is the use of the therapy control for the treatment of CHD, which is played out via the iATROS medical device. At the start of the digital treatment, the patients receive suitable measuring devices for recording their vital parameters in the home environment. With the completion of the visit in month 9, the active phase of the study has ended. Patients will now use the iATROS medical device for another 9 months, after which the stability of the intervention effects will be determined.
  Interventions: Device: CHD therapy through iATROS medical device
- Group without the medical device "iATROS": All patients in the control group will receive standard-of-care treatment in the 9 months after randomization. There will be no further intervention during this phase. Similarly, treatment is not influenced or restricted in terms of free choice of medical care or medical treatment.
  Subsequently, they also receive access to the iATROS medical device. Patients will receive suitable measuring devices for recording their vital parameters in the home environment. The effects of the intervention will be recorded after 9 months.

INTERVENTIONS:
Device: CHD therapy through iATROS medical device — The intervention to be carried out in the treatment group is the use of the therapy control for the treatment of CHD played out via the iATROS medicine product. Patients will receive a suitable and medical device certified measuring device for recording vital parameters. The iATROS app is downloaded to the patient's smartphone and the app is activated by entering a code that identifies the user as a participant in the study. When using the app for the first time, the patient is guided through the first steps of using the app and asked to transfer his or her health data to the app. The therapy control by means of the medication product takes place over the entire duration of the study.
  Groups: Group with the medical device "iATROS"

SUMMARY:
This study will test a controlled investigation of the efficacy and effectiveness of iATROS digital therapy management for risk factor adjustment in patients with coronary heart disease (CHD).

DETAILED DESCRIPTION:
The purpose of this study is to determine the efficacy and effectiveness of iATROS digital therapy management for risk factor adjustment in patients with coronary heart disease compared to the medical standard of care.

In addition, data will be provided to investigate the functionality of the rule engine in the treatment of CHD patients and insights will be gained for the further development of this component of the iATROS platform for the digital and intelligent treatment of patients.

Furthermore, the use of digital everyday products (smartphones) in secondary prevention and therapy management of CHD patients will be considered.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years
* Patients diagnosed with ischemic heart disease according to ICD I20 to I25 who also have at least one of the following:

  1. inpatient stay with acute STEMI/NSTEMI or historic STEMI/NSTEMI; and/or
  2. Coronary stent implantation, angioplasty or bypass surgery that has taken place.
* Ownership and use of a smartphone that allows installation and use of "iATROS," where "use" requires having the physical and mental ability to use and apply the iATROS app.
* Insured with the cooperating insurances

Exclusion Criteria:

* No use of a smartphone
* Lack of the linguistic, physical and mental abilities necessary to use the iATROS app, or to use so-called "apps" on a smartphone or tablet in general.
* Absolute contraindications: Any disease associated with a reduced life expectancy of less than 2 years; Any disease/condition that limits participation in the program; Pregnant or breast feeding patients; Patients with advanced dementia
* Existing participation and enrollment in an iATROS health program.
* Participation in another clinical trial if participation results in complications with compliance, measures to be performed, bias of results, or status of treatment according to the current standard of care.
* Comorbidities or the presence of another physical condition that complicates the setting of the clinical target parameters sought in the study (i.e., if, due to the patient's individual situation, a different value would have to be issued as the target value for a clinical parameter to be classified as healthy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult (≥ 18 years) patients with a diagnosis of coronary artery disease at study inclusion AND one of the following conditions: Diagnosis of STEMI/NSTEMI , OR they have had coronary intervention (eg, stent, angioplasty, or bypass surgery) or a similar formulation, are eligible to participate in the study as long as they meet the inclusion/exclusion criteria and are insured by the cooperating insurers.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-10-05 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients in target range of LDL or blood pressure | 9 months
  Proportion of patients per study arm in percent with adjusted LDL cholesterol in the blood of < 55 mg/dl (< 1.4 mmol/l) and/or adjusted blood pressure according to ESC guideline (≤130 mmHg systolic or ≤140 mmHg systolic for age > 70 years).

SECONDARY OUTCOMES:
Absolute LDL reduction after 9 months in patients with known LDL levels at inclusion (not older than 12 months at study inclusion) and no medication adjustment within the last 12 months prior to study inclusion. | 9 months
  Comparison of the mean value of the absolute reduction between the treatment and control group of this patient population with regard to statistically significant differences.
  Furthermore, intra-group comparison of this patient population per study arm to determine statistically significant effects with regard to LDL reduction by treatment with iATROS over 9 months.
Assessment of stability: Comparison of LDL levels after 18 months in patients with known LDL levels | 18 months
  Comparison of medical parameter LDL (available through standard-of-care treatment) between the two study arms after 18 months study duration.
Assessment of stability: Comparison of blood pressure after 18 months | 18 months
  Comparison of blood pressure values (available through standard-of-care measurements) between the two study arms after 18 months study duration.
In patients with diabetes: target blood HbA1c level of ≤ 7% or ≤ 53mmol/mol after 9 months. | 9 months
  Comparison of the proportion of patients per study arm in percent in the HbA1c target range with regard to statistically significant differences. In addition to an intergroup comparison, an intragroup comparison per study arm will be performed.
Assessment of stability in patients with diabetes: Comparison of blood HbA1c levels after 18 months. | 18 months
  Comparison of medical parameter HbA1c (available through standard-of-care treatment) between the two study arms after 18 months study duration.
In patients with diabetes: absolute reduction in blood HbA1c level after 9 months. | 9 months
  Comparison of the mean absolute reduction in HbA1 levels between the treatment and control groups for statistically significant differences in patients with history of HbA1c levels at inclusion.
  Furthermore, intragroup comparison per study arm to determine, whether treatment with iATROS has a statistically significant effect on the reduction of HbA1c levels over 9 months.
In patients with obesity: absolute BMI reduction after 9 months. | 9 months
  Comparison of the mean value of the absolute BMI reduction and the absolute weight reduction in [kg] with regard to the statistical significance of the absolute change between all patients in the treatment and control group. In addition to an intergroup comparison, an intragroup comparison per study arm will be performed.
Assessment of stability in patients with obesity: Comparison of BMI changes after 18 months. | 18 months
  Comparison of BMI values (available through standard-of-care measurement of weight and height which will be combined to report BMI in kg/m^2) between the two study arms after 18 months study duration.
Absolute BMI reduction in patients with initial BMI > 30kg/m2 after 9 months. | 9 months
  Comparison of the mean value of the absolute BMI reduction of this patient collective as well as the mean absolute weight reduction in [kg] with regard to statistical significance of the absolute change between the treatment and the control group. In addition to an intergroup comparison, an intragroup comparison per study arm will be performed.
In patients with obesity: percentage reduction in body mass index (BMI) after 9 months, which should fall within the target range below 25 kg/m2 as best as possible according to guideline recommendations. | 9 months
  Comparison of the mean value of the percentage BMI reduction between the treatment and control groups with regard to statistical significance. In addition, a comparison with the predefined target value is to be used to calculate which proportion of the intervention and control groups falls within this target range in [%] before the study period and after 9 months. In addition to an intragroup comparison, an intragroup comparison per study arm will be performed.
For patients with current nicotine abuse: determination of/review of smoking cessation after 9 months. | 9 months
  Query of smoking status and pack years per patient. Comparison of the percentage per study arm, who no longer define themselves as "smokers" and the percentage of patients who have defined themselves as "ex-smokers" for >6 months. Comparison of study arms and intragroup comparison 9 months after inclusion.
  Determination of smoking status using the Fagerström test for nicotine dependence (FTND).
Assessment of stability for patients with current nicotine abuse: determination of/review of smoking cessation after 18 months. | 18 months
  Comparison of Fagerström test for nicotine dependence (FTND) scores between the two study arms after 18 months study duration.
Improving health literacy | 9 months and 18 months
  The study will examine whether an improvement in health literacy can be measured after 9 and 18 months when using digital therapy management via iATROS. The Rasch-scaled short form of the European Health Literacy Survey (HLS-EU-Q16) questionnaire comprises 16 questions that are rated on a 4-level scale, with the answer options focussing on the respective difficulty (very easy, fairly easy, fairly difficult, very difficult). The four answer options are dichotomised, whereby the two categories "very easy" and "fairly easy" were assigned a value of 1 and the two remaining categories a value of 0. Based on the sums achieved, the health literacy of the patients is finally categorised as "insufficient" (sum 0-8), "problematic" (sum 9-12) and "sufficient" (sum 13-16).Since the questionnaires are submitted in the treatment group and the control group both at baseline and after 9 and 18 months, respectively, an intra-group comparison as well as an inter-group comparison is possible.
Assessment of stability: Improving health literacy | 18 months
  Comparison of the European Health Literacy Survey (HLS-EU-Q16) scores between the two study arms after 18 months study duration.
Improving patient sovereignty | 9 months and 18 months
  The study will examine whether the use of iATROS results in an increase in patient sovereignty after the treatment period of 9 and also 18 months. In order to measure this, a short-form of the Patient Activation Measure (PAM-13) will be used. The results are divided into different categories by quantitatively evaluating the results of the questions answered in a four-point Likert scale (not true, hardly true, rather true, exactly true). The total score results from the answers to the individual questions after standardization and is divided into four levels: Level 1 (lack of belief that activation is important, ≤47 points), Level 2 (lack of knowledge and confidence to take action, 47.1-55.1 points), Level 3 (beginning to take action, 55.2-67.0 points) and Level 4 (taking action, ≥67 points). The measurement of PAM-13 at the beginning of the study and after 9 and 18 months allows an intragroup and intergroup comparison.
Assessment of stability: Improving patient sovereignty | 18 months
  Comparison of the Patient Activation Measure (PAM-13) scores between the two study arms after 18 months study duration.

CONTACTS AND LOCATIONS:
Overall Officials: Moritz Sinner, PD Dr. med, Principal Investigator — Medizinische Klinik I und Poliklinik LMU Klinikum Campus Großhadern; Stefan Kääb, Prof.Dr.med., Principal Investigator — Medizinische Klinik I und Poliklinik LMU Klinikum Campus Großhadern
Locations (1):
- Klinikum der Ludwig-Maximilians-Universität München (Klinikum der Universität München), Medizinische Klinik und Poliklinik I, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No